CLINICAL TRIAL: NCT00196326
Title: A Multicenter, Open-label Study to Evaluate the Efficacy and Safety of an Extended-cycle, Low Dose, Combination Oral Contraceptive, Which Utilizes Ethinyl Estradiol During the Seven Day Interval Between Each 84-day Cycle
Brief Title: Open-label Study to Evaluate the Efficacy and Safety of an Extended-cycle, Low Dose Combination Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Druamed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DR-PSE-309
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2009-04-15 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: Contraception
Keywords: pregnancy prevention; oral contraceptives
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DR-1011 (Experimental): Participants were instructed to take, by mouth, one tablet daily for four 91-day cycles.
  Interventions: Drug: DR-1011

INTERVENTIONS:
Drug: DR-1011 — Eighty-four orange, embossed tablets, each containing 100 μg levonorgestrel (LNG) / 20 μg ethinyl estradiol (EE) and 7 yellow, embossed tablets, each containing 10 μg of EE. One combination tablet was to be taken each day for 84 days followed by 7 days of EE tablets in 91-day cycles repeated consecutively for approximately one year (four 91-day cycles).
  Other Names: levonorgestrel/ethinyl estradiol

SUMMARY:
This is an open-label, single treatment study. All subjects will receive one year of oral contraceptive therapy with DR-1011. Study participants will receive physical and gynecological exams, including Pap smear. During the study, all participants will be required to complete a diary.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Not pregnant or breastfeeding
* Sexually active at risk of pregnancy

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy within the last 3 months
* Smoking > 10 cigarettes per day

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2235 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (49):
- United States (49):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, New London, Connecticut
  - Duramed Investigational Site, Coral Cables, Florida
  - Duramed Investigational Site, Hollywood, Florida
  - Duramed Investigational Site, Jacksonville, Florida
  - Duramed Investigational Site, Leesburg, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Palm Springs, Florida
  - Duramed Investigational Site, Sarasota, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Douglasville, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Shawnee Mission, Kansas
  - Duramed Investigational Site, Topeka, Kansas
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Kansas City, Missouri
  - Duramed Investigational Site, St Louis, Missouri
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, New Brunswick, New Jersey
  - Duramed Investigational Site, Rochester, New York
  - Duramed Investigational Site, Charlotte, North Carolina
  - Duramed Investigational Site, Wilmington, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Willow Grove, Pennsylvania
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Waco, Texas
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Newport News, Virginia
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Richmond, Virginia
  - Duramed Investigational Site, Lakewood, Washington
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington

REFERENCES:
- [Result] Kroll R, Reape KZ, Margolis M. The efficacy and safety of a low-dose, 91-day, extended-regimen oral contraceptive with continuous ethinyl estradiol. Contraception. 2010 Jan;81(1):41-8. doi: 10.1016/j.contraception.2009.07.003. PMID 20004272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2968 subjects were screened and 2235 subjects were enrolled in the study. Of those enrolled, 2185 took at least one dose of study medication.
Period: Overall Study
Arm/Group | DR-1011
Started | 2235 (Took at least one dose of study medication)
Safety Population | 2185 (Treated participants)
Pregnancy Intent-to-treat Cohort (PITT) | 1735 (Completed one cycle and 18-35 years old)
Completed | 1249
Not Completed | 986
Not completed — Did not meet protocol requirements | 64
Not completed — Non-compliance with the protocol | 81
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 225
Not completed — Adverse Event | 253
Not completed — Pregnancy | 34
Not completed — Lost to Follow-up | 304
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | DR-1011
Number analyzed (Participants) | 2185
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2185
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 256
  Asian | 36
  Caucasian | 1627
  Hispanic | 218
  Other | 48
Region of Enrollment [Number; unit: participants]
  United States | 2185
Weight [Mean (Standard Deviation); unit: pounds] | 158.7 (41.26)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — n=2183
  kg/m^2 | 26.7 (6.65)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Pregnancy Rate (Pearl Index) For 91-Day Cycles by Cohort Using up to 14 Days Post-Last Combination Dose When Defining "On Drug" Pregnancy
Description: Pearl Index= ((100)*(number of pregnancies)*(4 cycles/year))/number of 91-day cycles completed.
  The pregnancy rate included "on-drug" pregnancies, defined as those pregnancies for which the date of conception was on or after the date of first dose of study medication, but no more than 14 days after the date of last combination dose of study medication.
  Pregnancy was defined as a positive pregnancy test verified by the study staff. The conception date was based on the ultrasound date. A pregnancy was not considered 'on drug' if conception clearly occurred prior to first dose of study medication, or more than 14 days after the date of last combination dose of study medication.
  Three denominators are reported;
  * excluding cycles where other birth control methods (BCMs) was used
  * all complete cycles
  * compliant-use (i.e. subject did not skip two or more consecutive pills or had a pattern of substantial non-compliance, or used a prohibited concomitant medication)
Time Frame: up to one year
Population: The pregnancy intent-to-treat cohort (PITT) consisted of subjects between the ages of 18 and 35 who were randomized to treatment and completed at least one cycle of study medication.
Measure: Number; unit: pregnancies per 100 woman years exposure
Arm/Group | DR-1011
Number analyzed (Participants) | 1735
pregnancies per 100 woman years exposure
  Excluding other BCMs (n=1732) | 2.44
  All complete cycles (n=1735) | 2.42
  Compliant-Use (n=1685) | 1.77

2. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: Safety was assessed by summarizing adverse events recorded in the patient's daily diary and reported by subjects at each study visit, and by summarizing results of examination, vital signs and clinical laboratory values.
Time Frame: Day 1 up to one year
Population: The safety cohort consisted of all patient who took at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | DR-1011
Number analyzed (Participants) | 2185
participants | 1742

3. Primary Outcome: Annualized Pregnancy Rate (Pearl Index) For 91-Day Cycles by Cohort Using up to 7 Days Post-Last Combination Dose When Defining "On Drug" Pregnancy
Description: Pearl Index= ((100)*(number of pregnancies)*(4 cycles/year))/number of 91-day cycles completed.
  The pregnancy rate included "on-drug" pregnancies, defined as those pregnancies for which the date of conception was on or after the date of first dose of study medication, but no more than 7 days after the date of last combination dose of study medication.
  Pregnancy was defined as a positive pregnancy test verified by the study staff. The conception date was based on the ultrasound date. A pregnancy was not considered 'on drug' if conception clearly occurred prior to first dose of study medication, or more than 7 days after the date of last combination dose of study medication.
  Three denominators are reported;
  * excluding cycles where other birth control methods (BCMs) was used
  * all complete cycles
  * compliant-use (i.e. subject did not skip two or more consecutive pills or had a pattern of substantial non-compliance, or used a prohibited concomitant medication)
Time Frame: up to one year
Population: as for outcome 1
Measure: Number; unit: pregnancies per 100 woman years exposure
Arm/Group | DR-1011
Number analyzed (Participants) | 1735
pregnancies per 100 woman years exposure
  Excluding other BCMs (n=1732) | 2.15
  All complete cycles (n=1735) | 2.12
  Compliant-Use (n=1685) | 1.77

ADVERSE EVENTS:
Time Frame: Day 1 up to one year
Arm/Group | DR-1011
Serious Adverse Events (participants affected / at risk) | 34/2185
Other Adverse Events (participants affected / at risk) | 1333/2185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-1011 (N=2185)
ABDOMINAL PAIN UPPER (General disorders) | 1 (1)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 4 (4)
APPENDICITIS (Infections and infestations) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
BILIARY DILATATION (Hepatobiliary disorders) | 1 (1)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 (1)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CLEFT PALATE REPAIR (Surgical and medical procedures) | 1 (1)
CONGENITAL GENITAL MALFORMATION MALE (Pregnancy, puerperium and perinatal conditions) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1)
DRUG ABUSER (Social circumstances) | 1 (1)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1)
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
WOUND DECOMPOSITION (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-1011 (N=2185)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 175 (268)
DYSMENORRHOEA (Reproductive system and breast disorders) | 250 (460)
HEADACHE (Nervous system disorders) | 732 (2495)
METRORRHAGIA (Reproductive system and breast disorders) | 183 (291)
NASOPHARYNGITIS (Infections and infestations) | 362 (528)
NAUSEA (Gastrointestinal disorders) | 190 (272)
SINUSITIS (Infections and infestations) | 157 (198)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 174 (223)
URINARY TRACT INFECTION (Infections and infestations) | 118 (147)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can (i) review results communications prior to public release and can embargo communications regarding trial results for a period of at least 60 days but no more than 180 days from the time submitted to the sponsor for review; and (ii) require in instances of a multi-center study, that a single PI not disclose study data until after the multi-center results are published, provided such results are published within eighteen (18) months of the conclusion of the study.